CLINICAL TRIAL: NCT02670057
Title: Sphenopalatine Ganglion Block to Treat Shoulder Pain During and/or After Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00619
Record Dates: First submitted 2016-01-21; First posted 2016-02-01 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Ipsilateral Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transnasal SPG block (Experimental)
  Interventions: Procedure: Transnasal SPG block

INTERVENTIONS:
Procedure: Transnasal SPG block

SUMMARY:
The purpose of this open label pilot study is to evaluate the utility of sphenopalatine ganglion (SPG) block to manage ipsilateral shoulder pain (ISP) during and/or after cesarean.

DETAILED DESCRIPTION:
Shoulder pain thought to be caused by blood and amniotic fluid irritation of the diaphragm and nerves that supply the shoulder, can occur during and/or after a cesarean. Investigators will consent 100 patients, and will enroll 10 patients who develop ISP and have a score of is >5/10 on the Verbal Analog pain Scale (VAS). Patients will be their own controls. Transnasal SPG block will be performed after childbirth, and and beginning at 20 minutes post treatment, the patient will be asked to rate their shoulder pain using the VAS a number of times.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean
* Presence of post-operative ISP, VAS >5/10
* American Society of Anesthesiologists Class 1 - 3.
* No allergy to lidocaine

Exclusion Criteria:

* American Society of Anesthesiologists Class 4 or 5.
* Allergy to lidocaine
* Nasal pathology (e.g., deviated septum)
* Patients who receive sedatives during cesarean
* Bleeding diathesis
* Any patient who the PI feels will be unable to comply with all protocol related procedures
* Shoulder pain prior to cesarean

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Reduction of shoulder pain measured using Verbal Analog pain Scale (VAS) | 90 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Grant, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States